CLINICAL TRIAL: NCT05585268
Title: Electronic Decision Support for Deprescribing in Patients on Hemodialysis: a Prospective, Controlled, Quality Improvement Study
Brief Title: Electronic Decision Support for Deprescribing in Patients on Hemodialysis
Acronym: MedSafer-HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Emily McDonald, Associate Professor of Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0000
Record Dates: First submitted 2022-10-02; First posted 2022-10-18 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: End Stage Renal Disease; Hypertension; Diabete Type 2; Renal Failure Chronic; Anemia; Medication Interaction
MeSH Terms: conditions — Kidney Failure, Chronic; Hypertension; Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic; Anemia

STUDY DESIGN:
Intervention Model Description: This quality improvement, parallel group, superiority trial will use two different dialysis sites of the McGill University Health Centre. One unit will act as a control unit. The other will act as an intervention unit. Participants are automatically enrolled in the study and assigned to the intervention when the MedSafer reports are handed to the clinical team at the time of performing a medication reconciliation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MedSafer-supplemented medication reconciliation (Active Comparator): This unit will act as an intervention unit for the MedRec where MedSafer deprescribing reports will be handed to the treating team and deprescribing brochures from the Canadian Deprescribing Network will be given to patients.
  Interventions: Other: Medication reconciliation supplemented with MedSafer and deprescribing brochures
- Standard of care medication reconciliation (No Intervention): This unit will serve as the control unit where standard of care will be provided and no deprescribing reports nor brochures will be delivered. MedSafer reports will be generated but withheld from the clinical team. This will serve as a comparator to determine if the intervention unit was more successful in deprescribing compared to this control unit.

INTERVENTIONS:
Other: Medication reconciliation supplemented with MedSafer and deprescribing brochures — This unit will act as an intervention unit for the MedRec where MedSafer deprescribing reports will be handed to the treating team and deprescribing brochures from the Canadian Deprescribing Network will be given to patients.
  Arms: MedSafer-supplemented medication reconciliation

SUMMARY:
Dialysis patients are prescribed an average of 10-12 medications per day, from up to 4-5 different clinicians and have the heaviest pill burden of all chronic conditions given their degree of comorbidity. One strategy for addressing the problem of "medication overload" is through scalable deprescribing interventions. MedSafer is an electronic deprescribing tool that cross-references patient health data with existing deprescribing guidelines and provides a deprescribing report to clinicians to facilitate deprescribing and reducing the burden of polypharmacy. In this study the investigators will test MedSafer on dialysis patients paired with medication reconciliation on an intervention unit compared to a control unit.

DETAILED DESCRIPTION:
Patients on dialysis are prescribed an average of 10-12 medications per day from up to 4-5 different clinicians and amounting to up to 19 pills per day. This patient population has one of the the heaviest pill burdens of all chronic conditions because of therapy to treat comorbidities like disease, hypertension, or diabetes as well as therapy directed at symptoms and drug side effects.

Over 90% of hemodialysis patients take 5 or more medications (polypharmacy), contributing to medication overload. Further, up to 50% of patients on dialysis are prescribed a potentially inappropriate medication (PIM), defined as a medication carrying an increased risk of contributing to an adverse drug event (ADE). Polypharmacy and associated ADEs increase emergency room visits, hospital admissions and the risk of premature death. Furthermore, some medications have little therapeutic benefit and simply add to pill burden.

Studies continue to document the pressing need for deprescribing, medication reconciliation, and medication management programs in dialysis patient populations for the above reasons. While deprescribing guidelines are available to clinicians, they can be difficult to implement as few tools consolidate the recommendations, guidelines are often long lists which require memorization, and they may not explain how to deprescribe and what rebound symptoms to watch out for. The investigators have previously demonstrated that the electronic tool MedSafer, which identifies deprescribing opportunities based on comparing medication lists and comorbidities to a curated ruleset which incorporates publicly available deprescribing guidance and emerging literature, can be a valuable aid in supporting deprescription of PIMs during acute care episodes. MedSafer has also been shown to be of benefit in Long Term Care settings. Dialysis patients, with a large burden of polypharmacy and complex medical histories, coupled with a high risk for adverse drug events leading to hospitalization and death, represent a unique population in which to study a systematic deprescribing intervention as a means of improving quality of care.

Objectives The primary aim is to provide deprescribing reports containing MedSafer recommendations to the clinical team of a hemodialysis unit during the process of Medication reconciliation, to determine if the identification of deprescribing opportunities can improve medication appropriateness as defined by the receipt of potentially inappropriate medications (PIMs) at the patient level. This intervention will be compared to the efficacy of the intervention with a control dialysis unit that will undergo the standard of care medication reconciliation process with a MedSafer report.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* On outpatient maintenance hemodialysis
* On one of the study units

Exclusion Criteria:

* Patient is hospitalized during the period of the intervention
* Patient is newly initiated on hemodialysis during the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with one or more PIMs deprescribed | 1 month
  The proportion of participants with one or more PIMs deprescribed following a medication reconciliation, compared between intervention and control units.This will be conditioned on patients with 1 or more PIMs at baseline.

SECONDARY OUTCOMES:
Mean number of total medications | 1 month
  The reduction in the mean number of drugs taken following a medication reconciliation compared between intervention and control unit

CONTACTS AND LOCATIONS:
Overall Officials: Emily McDonald, MD MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymous data will be made available for secondary analysis upon request with a data sharing agreement
Supporting Information: Study Protocol, CSR
Time Frame: 1-year after publication of the main trial
Access Criteria: Contact the primary investigator at emily.mcdonald@mcgill.ca; a data sharing agreement will need to be in place.

REFERENCES:
- [Background] Marin JG, Beresford L, Lo C, Pai A, Espino-Hernandez G, Beaulieu M. Prescription Patterns in Dialysis Patients: Differences Between Hemodialysis and Peritoneal Dialysis Patients and Opportunities for Deprescription. Can J Kidney Health Dis. 2020 May 1;7:2054358120912652. doi: 10.1177/2054358120912652. eCollection 2020. PMID 32426145
- [Background] Moryousef J, Bortolussi-Courval E, Podymow T, Lee TC, Trinh E, McDonald EG. Deprescribing Opportunities for Hospitalized Patients With End-Stage Kidney Disease on Hemodialysis: A Secondary Analysis of the MedSafer Cluster Randomized Controlled Trial. Can J Kidney Health Dis. 2022 May 13;9:20543581221098778. doi: 10.1177/20543581221098778. eCollection 2022. PMID 35586025
- [Background] Battistella M, Jandoc R, Ng JY, McArthur E, Garg AX. A Province-wide, Cross-sectional Study of Demographics and Medication Use of Patients in Hemodialysis Units Across Ontario. Can J Kidney Health Dis. 2018 Mar 13;5:2054358118760832. doi: 10.1177/2054358118760832. eCollection 2018. PMID 29568537
- [Background] Alshamrani M, Almalki A, Qureshi M, Yusuf O, Ismail S. Polypharmacy and Medication-Related Problems in Hemodialysis Patients: A Call for Deprescribing. Pharmacy (Basel). 2018 Jul 25;6(3):76. doi: 10.3390/pharmacy6030076. PMID 30046021
- [Background] Sommer J, Seeling A, Rupprecht H. Adverse Drug Events in Patients with Chronic Kidney Disease Associated with Multiple Drug Interactions and Polypharmacy. Drugs Aging. 2020 May;37(5):359-372. doi: 10.1007/s40266-020-00747-0. PMID 32056163
- [Background] Halli-Tierney AD, Scarbrough C, Carroll D. Polypharmacy: Evaluating Risks and Deprescribing. Am Fam Physician. 2019 Jul 1;100(1):32-38. PMID 31259501
- [Background] Hovstadius B, Petersson G. Factors leading to excessive polypharmacy. Clin Geriatr Med. 2012 May;28(2):159-72. doi: 10.1016/j.cger.2012.01.001. Epub 2012 Feb 15. PMID 22500536
- [Background] McDonald EG, Wu PE, Rashidi B, Wilson MG, Bortolussi-Courval E, Atique A, Battu K, Bonnici A, Elsayed S, Wilson AG, Papillon-Ferland L, Pilote L, Porter S, Murphy J, Ross SB, Shiu J, Tamblyn R, Whitty R, Xu J, Fabreau G, Haddad T, Palepu A, Khan N, McAlister FA, Downar J, Huang AR, MacMillan TE, Cavalcanti RB, Lee TC. The MedSafer Study-Electronic Decision Support for Deprescribing in Hospitalized Older Adults: A Cluster Randomized Clinical Trial. JAMA Intern Med. 2022 Mar 1;182(3):265-273. doi: 10.1001/jamainternmed.2021.7429. PMID 35040926
- [Background] Nadeau ME, Henry JL, Lee TC, Bortolussi-Courval E, Goodine C, McDonald EG. Spread and scale of an electronic deprescribing software to improve health outcomes of older adults living in nursing homes: study protocol for a stepped wedge cluster randomized trial. Trials. 2021 Nov 2;22(1):763. doi: 10.1186/s13063-021-05729-0. PMID 34727956
- [Background] McDonald EG, Wu PE, Rashidi B, Forster AJ, Huang A, Pilote L, Papillon-Ferland L, Bonnici A, Tamblyn R, Whitty R, Porter S, Battu K, Downar J, Lee TC. The MedSafer Study: A Controlled Trial of an Electronic Decision Support Tool for Deprescribing in Acute Care. J Am Geriatr Soc. 2019 Sep;67(9):1843-1850. doi: 10.1111/jgs.16040. Epub 2019 Jun 27. PMID 31250427
- [Background] McIntyre C, McQuillan R, Bell C, Battistella M. Targeted Deprescribing in an Outpatient Hemodialysis Unit: A Quality Improvement Study to Decrease Polypharmacy. Am J Kidney Dis. 2017 Nov;70(5):611-618. doi: 10.1053/j.ajkd.2017.02.374. Epub 2017 Apr 14. PMID 28416321
- [Derived] Bortolussi-Courval E, Podymow T, Trinh E, Moryousef J, Hanula R, Huon JF, Mavrakanas T, Suri R, Lee TC, McDonald EG. Electronic Decision Support for Deprescribing in Patients on Hemodialysis: Clinical Research Protocol for a Prospective, Controlled, Quality Improvement Study. Can J Kidney Health Dis. 2023 Jun 26;10:20543581231165712. doi: 10.1177/20543581231165712. eCollection 2023. PMID 37435299